CLINICAL TRIAL: NCT01890174
Title: Repeatability and Reproducibility of Cirrus HD-OCT Macular Retinal Pigment Epithelium Elevation
Status: Completed | Type: Observational
Sponsor: Carl Zeiss Meditec, Inc. (Industry)
Collaborators: DataMed Devices Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HD-OCT-DR-2010-2
Record Dates: First submitted 2013-06-24; First posted 2013-07-01 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Dry AMD With Macular Drusen

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- AMD with macular drusen: Patients diagnosed with dry AMD with macular drusen

SUMMARY:
The objective of this study is to determine the repeatability and reproducibility of the Cirrus HD-OCT measurements of drusen area and volume.

DETAILED DESCRIPTION:
This is a prospective, single site study. Ocular history and examination will be conducted on consented subjects to determine further participation in the study. The study will be divided into two phases. In Phase 1, the inter-device variability of Cirrus HD-OCT measurements of drusen area and volume will be determined. In Phase 2, the inter-operator variability of Cirrus HD-OCT measurements of drusen area and volume will be determined. In each of these phases, the Macular Cube 200 x 200 scan and the Macular Cube 512 x 128 scan will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 50 years of age or older diagnosed to have dry AMD with macular drusen.
2. Drusen should not be combined with other lesions such as geographic atrophy (GA) or choroidal neovascularization.
3. Able and willing to make the required study visits.
4. Able and willing to give consent and follow study instructions.

Exclusion Criteria:

1. History of retinal surgery, laser photocoagulation, and/or radiation therapy to the eye.
2. Evidence of other retinal diseases of the eye, including wet AMD, diabetic retinopathy, diabetic macular edema, or significant vitreomacular traction.
3. Thick media opacity or inability to fixate that precludes obtaining acceptable scans.
4. Concomitant use of hydrochloroquine or chloroquine.
5. Unable to make the required study visits.
6. Unable to give consent or follow study instructions.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2011-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Coefficient of variation for area (mm^2) of RPE elevation measurements in the central 3 mm circle. | Single visit observation

SECONDARY OUTCOMES:
Coefficient of variation for volume (mm^3) of RPE elevation measurements in the central 3 mm circle. | Single visit observation

OTHER OUTCOMES:
Coefficient of variation for area (mm^2) of RPE elevation measurements in the central 5 mm circle. | Single visit observation
Coefficient of variation for volume (mm^3) of RPE elevation measurements in the central 5 mm circle. | Single visit observation

CONTACTS AND LOCATIONS:
Overall Officials: Mark Wieland, MD, Principal Investigator — Northern California Retina Vitreous Associates Medical Group, Inc.
Locations (1):
- Northern California Retina Vitreous Associates, Mountain View, California, United States

REFERENCES:
- [Background] Schmitz-Valckenberg S, Fleckenstein M, Scholl HP, Holz FG. Fundus autofluorescence and progression of age-related macular degeneration. Surv Ophthalmol. 2009 Jan-Feb;54(1):96-117. doi: 10.1016/j.survophthal.2008.10.004. PMID 19171212